CLINICAL TRIAL: NCT03276312
Title: Local Inoculation of Autologous Micro-fragmented Adipose Tissue in the Treatment of Minor Amputations of Diabetic Foot: A Randomized Controlled Trial
Brief Title: Autologous Micro-fragmented Adipose Tissue in the Treatment of Minor Amputations of Diabetic Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Giulia Trevisi Borsari, Dr, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADF01
Record Dates: First submitted 2017-07-24; First posted 2017-09-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Foot
Keywords: Lipogems; Adipose-derived Mesenchymal Stem Cells; Lipofilling; Diabetic foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Lipogems - local injection of autologous micro-fragmented adipose tissue
  Interventions: Device: Lipogems
- Control (No Intervention): Routine clinical practice

INTERVENTIONS:
Device: Lipogems — Lipogems® is an innovative system that, starting from minimum quantities of autologous lipoaspirate, provides, with a minimal manipulation, a micro-fragmented and non-expanded adipose tissue product
  Arms: Intervention

SUMMARY:
This is a randomized controlled monocentric study on 114 diabetic patients with the aim of evaluating the efficacy of the lipofilling with Lipogems® system in diabetic patients that are candidates for a minor amputation in the foot. In particular, it will be evaluated whether the lipofilling will be able to shorten the healing times and to reduce the number of major amputations, with consequent positive impact on the quality of life. Patients will be randomized to the treatment group with Lipogems® (local injection of autologous micro-fractured adipose tissue) or to the control group, thus, treatment according to standard clinical practice.

DETAILED DESCRIPTION:
Primary objective of this study is the evaluation of the time of the healing of the lesions resulting from minor amputations (digital or forefoot) treated with Lipogems® technique.

Secondary objectives are: 1) assessment of the safety of the lipofilling; 2) evaluation of the intensity of pain (VAS); 3) assessment of the skin tropism; 4) calculation of the relapse rate (defined as the occurrence of local infections, dehiscence and suffering of skin flaps that lead to a revision of the amputation stump or amputation at a higher level); 5) evaluation of the time of hospitalization and quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diabetes (diabetes mellitus type 1 and type 2) of both sexes over the age of 18 years.
2. Presence of irreversible gangrene digital or localized at forefoot (with X-ray of the foot negative or positive for osteolytic lesions at phalanges and/or metatarsus).
3. Patients with vascular problems absent or resolved (evaluated with Eco Color Doppler and ABI (Ankle Brachial Index, that calculates the ratio of the systolic pressure measured at the ankle and the systolic pressure in the arm, both measured in supine position using wave continue Doppler. If assessable, it has to be greater than/equal to 0.7) and pressure index finger/arm TBI (Toe Brachial Index, if assessable, it has to be greater than/equal to 0.6) and/or by the determination of the transcutaneous oxygen pressure (TcPO2 that needs to be equal to or greater than 30mmHg).

Exclusion Criteria:

1. Oncological treatments ongoing or previous (past 5 years) and/or neoplastic lesions
2. Patient under steroid therapy
3. Active vascular issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Healing time | 6 months
  Healing time after the minor amputation intended as the complete healing of the amputation stump

SECONDARY OUTCOMES:
Safety: All types of adverse events will be collected | 6 months
  All types of adverse events will be collected
Incidence of relapse | 6 months
  Relapse is intended as revision of the amputation stump or amputation at a higher level
Pain assessed using the Visual Analogue Scale (VAS) for pain | 6 months
  Pain will be assessed using the VAS pain scale
Total time of hospitalization | 6 months
  Hospitalization of the patient will be assessed counting the number of days in hospital
Total time of immobility | 6 months
  Immobility of the patient will be assessed counting the number of bed rest days
Quality of Life using the Short Form 36 (SF-36) questionnaire | 6 months
  Assessment of the quality of life (QoL) before surgery and during all the subsequent follow up visits using the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Silingardi, Prof, Principal Investigator — Baggiovara Hospital, Vascular Surgery department
Locations (1):
- University of Modena and Reggio Emilia, Modena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gennai S, Leone N, Covic T, Migliari M, Lonardi R, Silingardi R. Health-related quality of life outcomes and hospitalization length of stay after micro-fragmented autologous adipose tissue injection in minor amputations for diabetic foot ulceration (MiFrAADiF Trial): results from a randomized controlled single-center clinical trial. Int Angiol. 2021 Dec;40(6):512-519. doi: 10.23736/S0392-9590.21.04570-3. Epub 2021 Sep 13. PMID 34515448
- [Derived] Lonardi R, Leone N, Gennai S, Trevisi Borsari G, Covic T, Silingardi R. Autologous micro-fragmented adipose tissue for the treatment of diabetic foot minor amputations: a randomized controlled single-center clinical trial (MiFrAADiF). Stem Cell Res Ther. 2019 Jul 29;10(1):223. doi: 10.1186/s13287-019-1328-4. PMID 31358046